CLINICAL TRIAL: NCT02567396
Title: A Phase I Study of Single Agent Talazoparib (BMN 673) in Advanced Cancer Patients With Hepatic and Renal Dysfunction
Brief Title: Talazoparib in Treating Patients With Advanced or Metastatic Solid Tumors That Cannot Be Removed by Surgery and Liver or Kidney Dysfunction
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Other- Protocol moved to Disapproved
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-01641; NCI-2015-01641 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PJC-022; PJC-022 (Other: University Health Network Princess Margaret Cancer Center LAO); 9942 (Other: CTEP); UM1CA186644 (NIH)
Record Dates: First submitted 2015-10-02; First posted 2015-10-05 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Estrogen Receptor Negative; Head and Neck Squamous Cell Carcinoma; HER2/Neu Negative; Hormone-Resistant Prostate Cancer; Metastatic Pancreatic Adenocarcinoma; Progesterone Receptor Negative; Solid Neoplasm; Stage III Mesothelioma; Stage IIIA Gastric Cancer; Stage IIIA Non-Small Cell Lung Cancer; Stage IIIA Ovarian Cancer; Stage IIIA Small Cell Lung Carcinoma; Stage IIIB Gastric Cancer; Stage IIIB Non-Small Cell Lung Cancer; Stage IIIB Ovarian Cancer; Stage IIIB Small Cell Lung Carcinoma; Stage IIIC Gastric Cancer; Stage IIIC Ovarian Cancer; Stage IV Mesothelioma; Stage IV Non-Small Cell Lung Cancer; Stage IV Ovarian Cancer; Stage IV Small Cell Lung Carcinoma; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Mesothelioma; Stomach Neoplasms; Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms; Small Cell Lung Carcinoma; Triple Negative Breast Neoplasms | interventions — talazoparib

ARMS (1):
- Treatment (talazoparib) (Experimental): Patients receive talazoparib PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Talazoparib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Talazoparib — Given PO
  Other Names: BMN 673; BMN-673

SUMMARY:
This phase I trial studies the side effects and best dose of talazoparib in treating patients with solid tumors that have spread to other places in the body and usually cannot be cured or controlled with treatment (advanced) or have spread to other places in the body (metastatic) and cannot be removed by surgery and liver or kidney dysfunction. Talazoparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine safety, tolerability and recommended phase 2 dose (RP2D) of talazoparib in patients with varying degrees of hepatic and renal dysfunction.

SECONDARY OBJECTIVES:

I. To observe preliminary antitumor activity of talazoparib in patients with cancers that commonly harbor defects in homologous recombination repair.

II. To assess the pharmacokinetic (PK) profiles of talazoparib in patients with varying degrees of hepatic and renal dysfunction.

III. To evaluate the pharmacodynamic (PD) effects of talazoparib. IV. To evaluate biomarkers associated with response or resistance to talazoparib.

OUTLINE: This is a dose-escalation study. Patients are assigned to 1 of 6 cohorts based on the degree of hepatic or renal dysfunction.

Patients receive talazoparib orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* Any advanced solid malignancy will be eligible, with a strong preference for tumors that are known to commonly harbor defects in homologous recombination repair including triple-negative breast cancer, high-grade serous ovarian cancer, non-small cell lung cancer, small cell lung cancer, mesothelioma castration-resistant prostate cancer, pancreatic adenocarcinoma, gastric cancer and head & neck squamous cell cancer
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 criteria
* All patients must have completed any prior chemotherapy, targeted therapy, radiotherapy (unless palliative doses which must be discussed with study principal investigator), and surgery, >= 28 days before study entry
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 3 months
* Able to swallow and retain orally-administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 90 g/L
* Hepatic and renal function meeting the strata as outlined below; nota bene (NB): patients must fulfill both total bilirubin and serum glutamic-oxaloacetic transaminase (SGOT)/aspartate aminotransferase (AST) criteria and creatinine function to be included in a group; however, if a patient's total bilirubin and SGOT/AST and creatinine levels indicate different groups, the patient may be enrolled in the indicated group with the greatest degree of liver dysfunction; all liver and renal function tests must be completed within 24 hours prior to the start of treatment; Note: patients on dialysis will not be eligible

  * Group A: hepatic function: normal function (bilirubin =< upper limit of normal [ULN]; AST =< ULN); renal function: normal function (creatinine clearance [CrCl] >= 60 mL/min)
  * Group B: hepatic function: normal function (bilirubin =< ULN; AST =< ULN); renal function: moderate dysfunction (CrCl >= 30 and < 60 ml/min)
  * Group C: hepatic function: normal function (bilirubin =< ULN; AST =< ULN); renal function: severe dysfunction (CrCl >= 15 and < 30 ml/min)
  * Group D: hepatic function: mild dysfunction D1: bilirubin =< ULN; AST > ULN, D2: bilirubin > ULN and =< 1.5 x ULN; any AST; renal function: normal function (creatinine clearance [CrCl] >= 60 mL/min)
  * Group E: hepatic function: mooderate dysfunction (bilirubin 1.5 x > ULN and =< 3 x ULN; any AST); renal function: normal function (creatinine clearance [CrCl] >= 60 mL/min)
  * Group F: hepatic function: severe dysfunction (bilirubin > 3 x ULN and up to investigator's discretion; any AST); renal function: normal function (creatinine clearance [CrCl] >= 60 mL/min)
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of talazoparib administration
* All prior treatment-related toxicities must be Common Terminology Criteria for Adverse Events (CTCAE) v4.03 grade =< 1 (except for adverse events [AEs] not considered to be dose-limiting toxicities [DLTs] in this trial such as alopecia and lymphopenia) at the time of enrollment; if there are any questions, please contact the study's principal investigator
* Females of childbearing potential must have a negative serum pregnancy test at screening
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior treatment with talazoparib or a poly(adenosine diphosphate [ADP]-ribosyl)ation (PARP)1/2 inhibitor; prior treatment with other agents that inhibit deoxyribonucleic acid (DNA) repair (i.e. WEE1 homolog [S. pombe] [WEE1] inhibitors, ataxia telangiectasia mutated [ATM] inhibitors), is allowed; if there are any questions, please contact the study's principal investigator
* Any major surgery, extensive radiotherapy, chemotherapy with delayed toxicity, biologic therapy, or immunotherapy must not be given within 28 days prior to study enrollment; for daily or weekly chemotherapy without the potential for delayed toxicity, a washout period of 14 days prior to enrollment may be acceptable, and questions related to this can be discussed with study principal investigator
* Clinically significant bleeding diathesis or coagulopathy, including known platelet function disorders
* Known hypersensitivity to any of the components of talazoparib
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to talazoparib
* Use of other investigational drugs within 28 days (or five half-lives, whichever is shorter; with a minimum of 14 days from the last dose) preceding the first dose of talazoparib and during the study
* Symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression; patients with treated central nervous system (CNS) metastasis, no longer requiring steroid therapy are potentially eligible; patients with primary glioblastoma multiforme not requiring steroid therapy will be eligible
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, clinically significant cardiac arrhythmias, or psychiatric illness/social situations that would limit compliance with study requirements
* Any other known malignancy within 3 years (with the exception of non-melanoma skin cancer that had undergone curative treatment, cervical cancer in situ, or ductal/lobular carcinoma in situ of the breast that has underwent local treatment); consult the Cancer Therapy Evaluation Program (CTEP) medical monitor if unsure whether second malignancies meet the requirements specified above
* Women of childbearing potential should be advised to avoid pregnancy and use effective methods of contraception for 4 months after study treatment is completed; men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception for at least 4 months after study treatment is completed; if a female patient or a female partner of a patient becomes pregnant while the patient receives talazoparib, the potential hazard to the fetus should be explained to the patient and partner (as applicable)
* Active hepatitis B virus (HBV), or hepatitis C virus (HCV) infection (patients with chronic or cleared HBV and HCV infection are eligible)
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Any condition or medical problem in addition to the underlying malignancy and organ dysfunction that the investigator feels would pose unacceptable risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of toxicity, graded according to the National Cancer Institute (NCI) CTCAE version 4.03 | Up to 4 weeks after completion of study treatment
  Frequency and severity of adverse events will be tabulated using counts and proportions detailing frequently occurring, serious and severe events of interest. Adverse events will be summarized using all adverse events experienced, although a sub-analysis may be conducted including only those adverse events in which the treating physician deems possibly, probably or definitely attributable to study treatment.
Recommended phase 2 dose of talazoparib, graded according to NCI CTCAE version 4.0 | Up to 28 days
Tolerability of talazoparib in patients with varying degrees of hepatic and renal dysfunction | Up to 4 weeks after completion of study treatment

SECONDARY OUTCOMES:
Biomarkers associated with response or resistance to talazoparib | Up to 4 weeks after completion of study treatment
Objective response, graded according to RECIST version 1.1 | Up to 4 weeks after completion of study treatment
  If no objective responses are observed in a dose expansion cohort with a minimum of 10 patients evaluable for response, there is >= 89% probability to exclude a true objective response rate of >= 20%.
PK profiles of talazoparib in patients with varying degrees of hepatic and renal dysfunction | Pre-dose, and 30 minutes, 1, 2, 4, 6, 8, and 24 hours post-dose on day 1 of course 2, and pre-dose on day 1 of courses 3 and 4
  Attempts to model associations between pharmacokinetic data with toxicity profiles will be performed primarily using descriptive statistics; however, logistic regression may be used if warranted.
Progression-free survival (PFS) | Up to 4 weeks after completion of study treatment
  PFS will be investigated using logistic regression, Cox proportional hazards regression and/or generalized estimating equations as appropriate. Potential predictors include clinical predictors and molecular correlates. Descriptive statistics and plotting of data will also be used to better understand potential relationships.
Response rate | Up to 4 weeks after completion of study treatment
  Response rate will be investigated using logistic regression, Cox proportional hazards regression and/or generalized estimating equations as appropriate. Potential predictors include clinical predictors and molecular correlates. Descriptive statistics and plotting of data will also be used to better understand potential relationships.

OTHER OUTCOMES:
The pharmacodynamic effects of talazoparib | Up to day 2 of course 2

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Renouf, Principal Investigator — University Health Network Princess Margaret Cancer Center LAO